CLINICAL TRIAL: NCT04817891
Title: Cholinergic Functions and Modulation of the Cingulo-opercular Alertness Network in LBD
Brief Title: Stimulation of Cingulo-opercular Alertness Network
Acronym: SCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Benjamin Hampstead, PhD, Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00184296; R21AG069387 (NIH)
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Lewy Body Disease; Lewy Body Variant of Alzheimer Disease; Lewy Body Dementia With Behavioral Disturbance
Keywords: Lewy Body Dementia; Cognitive; Thinking; Cognition; Cognitive Rehabilitation; Brain Stimulation; Imaging; Lewy Body; Dementia
MeSH Terms: conditions — Lewy Body Disease; Lewy Body Variant of Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: Eligible participants receive individualized intervention/stimulation based on their fMRI and PET imaging.
Masking Description: Investigator, Outcomes Assessor, and Participant/Care Provider will all know the participant is receiving intervention/stimulation. There is no placebo condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Experimental: HD-tDCS (Experimental): Maximum 4 milliAmp (mA) per channel of HD-tDCS treatment for 20 minutes, for 10 sessions. Total mA dose determined by individualized computational models.
  Interventions: Device: HD-tDCS

INTERVENTIONS:
Device: HD-tDCS — Participants will receive HD-tDCS at up to 4 mA per channel for 20 minutes for 10 sessions. Dose determined through individualized computational models.

SUMMARY:
Fluctuations in alertness are very common in persons with Lewy body dementias and are a major source of disability. Changes in a chemical messenger molecule called acetylcholine within certain brain regions may play a role in these fluctuations. We propose to test this hypothesis and also determine whether a non-invasive way of stimulating affected brain regions may be of relevance for future management of these fluctuations.

DETAILED DESCRIPTION:
The central premise of the research study was that cholinergic system changes in specific neural network regions underlie cognitive fluctuations in patients with LBD. The cingulo-opercular task control (COTC) neural network is believed to play a role in maintenance of alertness but this remains uncertain in LDB. This critical knowledge gap formed the basis of the study's first aim. The study proposed to use transcranial direct current stimulation (tDCS) to "excite" critical cholinergic denervation components of the COTC as an adjunct to cholinergic pharmacotherapy in a target engagement study. tDCS is an emerging non-invasive neurostimulation technology that may improve a range of neurological symptoms, including cognition. The study evaluated whether target engagement by tDCS excitation of cholinergic denervated COTC hubs may affect cognitive fluctuations in LBD subjects.

While the cingulo-opercular network was expected to be the primary site of cholinergic denervation based on preliminary evidence, and thus the focus of the stimulation intervention, the typical pattern of cholinergic denervation in our sample occurred at a temporal lobe region that is classified as a node of the ventral attention network in the Gordon atlas. Additional results from examining different networks have been added to reflect the unanticipated relocation of stimulation location.

ELIGIBILITY:
Inclusion Criteria:

* LBD patients (DLB or PDD) who have cognitive fluctuations and who are on stable doses of cholinesterase inhibitors (i.e., at least 4 weeks) will be recruited to participate in this study.
* DLB patients will meet the Fourth consensus report of the DLB Consortium inclusion criteria for probable DLB.
* Subjects will be identified according to the following recognized DLB features: spontaneous parkinsonian motor signs, fluctuating attention and concentration, recurrent well-formed visual hallucinations, presence of REM behavioral sleep disturbance, anosmia/hyposmia,or autonomic dysfunction.
* PDD patients will meet the criteria by Emre et al. (Cognitive deficits in at least two of four of the following cognitive domains: Impaired attention, impaired executive functions, impairment in visuo-spatial functions, impaired free recall memory typically improved with cuing. Must also meet criteria for at least one behavioral symptom: apathy, depressed or anxious mood, hallucinations, delusions, excessive daytime sleepiness). Lack of behavioral symptoms does not exclude the diagnosis. Must also have none of Group III features present: (1) Co-existence of any other abnormality which might cause impairment, but judged not to be the cause of dementia. (2) Time interval between development of motor and cognitive symptoms not known. Must also have none of Group IV symptoms present: (1) Cognitive and behavioral symptoms appear solely in the context of other conditions such as acute confusion caused by systemic diseases or abnormalities, drug intoxication, or major depression according to DSM IV. (2) Features compatible with Probable Vascular Dementia criteria accordingly to NINDS-AIREN.

Exclusion Criteria:

* Subjects with contra-indications to MR imaging and/or tDCS, including pacemakers or claustrophobia
* Evidence of large vessel stroke or mass lesion on MRI
* Use of anti-cholinergic or neuroleptic drugs
* Evidence of atypical parkinsonism on neurological exam
* Major psychiatric illness, such as bipolar disorder
* Neurological conditions such as epilepsy, stroke, multiple sclerosis, or moderate to severe brain injury
* Sensory impairments that significantly limit one's ability to see or hear
* A significant history of recent alcohol or drug dependence
* Previous major radiation exposure
* Pregnancy

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Hampstead, PhD, Principal Investigator — University of Michigan
Locations (1):
- 4250 Plymouth Road (University of Michigan), Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled are those who consented to be in the study. They then underwent a screening process. Three participants did not continue after the screening process.
Groups:
- Experimental: HD-tDCS: HD-tDCS treatment for 20 minutes, repeated across 10 sessions (3-5 sessions/week). The pattern and dose of stimulation was individualized for each participant to generate electric field in regions of cholinergic denervation, as determined by reduced FEOBV binding. A maximum of 4 milliamps (mA) of current was delivered at each anode.
Period: Overall Study
Arm/Group | Experimental: HD-tDCS
Started | 15
Began Study Treatment (Participants who began treatment after consenting) | 13
Completed | 12
Not Completed | 3
Not completed — Did not pass screening after consenting to participate | 1
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Baseline is considered to be the participants who were deemed eligible to receive the study intervention (tDCS)
Arm/Group | Experimental: HD-tDCS
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] — Age is reported on the number of participants who were eligible to receive study intervention
  years | 75.77 (5.75)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex is reported on the number of participants who were eligible to receive study intervention
  Participants
    Female | 2
    Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity is reported on the number of participants who were eligible to receive study intervention
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 13
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race is reported on the number of participants who were eligible to receive study intervention
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 13
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Region of enrollment is reported on the number of participants who were eligible to receive study intervention
  participants
    United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Dementia Cognitive Fluctuations Scale
Description: Score on a 4-item subscale of the 17-item Dementia Cognitive Fluctuation Scale (DCFS), developed to address limitations in prior scales and has good test-retest and inter-rater reliability; this subscale highly discriminates between dementia with Lewy bodies (DLB) and other dementia groups. The DCFS is a subjective report of cognitive fluctuation, the spontaneous change in cognitive ability which is a core diagnostic feature of DLB. Total subscale scores range from 4 to 20, with higher scores indicating greater cognitive fluctuations. A decrease in score between Baseline and Post-Testing indicates an improvement in cognitive fluctuation.
Time Frame: Baseline and Post-Testing (3-4 weeks)
Population: Data is reported for participants who completed both baseline and week 3/4 measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: HD-tDCS
Number analyzed (Participants) | 12
score on a scale
  Baseline | 11.75 (3.31)
  Week 3/4 | 8.33 (1.56)
Statistical Analysis 1: Comparison: Experimental: HD-tDCS; Test type: Superiority; p < 0.001, t-test, 1 sided

2. Secondary Outcome: Resting State fMRI
Description: Functional connectivity measures whether activity in different brain regions show similar patterns of change over time. Graph theory metrics of resting-state fMRI can characterize functional connectivity among nodes (regions) of a brain network, and well as between nodes of different brain networks. Network segregation is the difference of within-network and between-network connectivity as a proportion of within-network connectivity, such that higher numbers reflect more segregation. Given that network segregation typically decreases with normal and pathological aging, higher network segregation is generally considered cognitively beneficial.
  Network segregation was examined for the ventral attention network (the actual focus of stimulation based on observed cholinergic denervation) and the original cingulo-opercular network, which was predicted at the time of grant proposal (but not supported by the observed cholinergic denervation).
Time Frame: Baseline and Post-Testing (3-4 weeks)
Population: Ten participants completed resting-State fMRI at Baseline and Post-Testing. Two participants were not eligible for MRI.
Measure: Mean (Standard Deviation); unit: ratio of network segregation
Arm/Group | Experimental: HD-tDCS
Number analyzed (Participants) | 10
ratio of network segregation
  Baseline - Ventral Attention Network | 0.23 (0.17)
  3/4 weeks - Ventral Attention Network | 0.33 (0.10)
  Baseline - Cingulo-opercular network | 0.53 (0.11)
  3/4 weeks - Cingulo-opercular network | 0.53 (0.11)
Statistical Analysis 1: Comparison: Experimental: HD-tDCS; Test type: Superiority; p = 0.018, t-test, 2 sided — p value for the Ventral Attention Network (network segregation)
Statistical Analysis 2: Comparison: Experimental: HD-tDCS; Test type: Superiority; p = 0.944, t-test, 2 sided — p value for the Cingulo Opercular Network (network segregation)

3. Secondary Outcome: Stroop Color Word Interference Test - Cognitive Control Performance
Description: Outcome Measure Description: Interference score in time to complete the Color Word Interference Test version of the Stroop task from the Delis-Kaplan Executive Function System. Participants 1) identify a series of colors, 2) read color words (e.g. blue) all written in black ink, and 3) name the ink color of color words printed in incongruous colored inks (e.g. for the word "green" written in red ink, the correct response is "red"). Tasks are performed as quickly as possible. Time to complete each task is recorded.
  Interference score is calculated as the time to complete the color-word (interference) test (CWT), less the average of the time to complete the color task (CT) and word-reading task (WT): CWT - ((CT + WT)/2). The score has a theoretical valid range of 0 - 300; a lower score suggests better cognitive control. A negative change (decrease) in score between Baseline and Post-Testing indicates improvement in cognitive control performance.
Time Frame: Baseline, 3-4 weeks
Population: 8 participants completed the Color Word Interference Test at Baseline and Post-Testing. 4 participants did not complete the test. Negative scores are technically possible, but given the known robust and reliable cognitive effort required in color word interference, a negative interference score would call into question the validity of the administration and be excluded. No participants' scores were negative and therefore none were excluded for this reason..
Measure: Mean (Standard Deviation); unit: calculated score
Groups:
- Experimental: HD-tDCS: HD-tDCS treatment for 20 minutes, repeated across 10 sessions (3-5 sessions/week). The pattern of stimulation was individualized for each participant to generate electric field in regions of cholinergic denervation, as determined by reduced FEOBV binding. A maximum of 4 milliamps of current was delivered at each anode.
Arm/Group | Experimental: HD-tDCS
Number analyzed (Participants) | 8
calculated score
  Baseline | 143.44 (51.89)
  3-4 weeks | 125.15 (52.91)
Statistical Analysis 1: Comparison: Experimental: HD-tDCS; Test type: Superiority; p = 0.239, t-test, 1 sided

4. Secondary Outcome: Objective Measures of Working Memory (N-back Test)
Description: The n-back test is a working memory task where a participant identify a stimulus that matches the stimulus experienced "n" steps back. Participants performed a 2-back test, in which they were asked to remember and press a button when presented with a stimulus that appeared two steps before the current one (e.g. square, circle, square).
  The number of correct and incorrect identifications are normalized (z-score). Total score is the z-score of correct button presses minus the z-score of incorrect button presses. Possible scores range from -4.85 to 4.85.
  A higher score (d') reflects better discrimination between target and non-target stimuli, and therefore better working memory performance. A positive change (increase) in 2-back score (d') between Baseline and Post-Testing indicates an improvement in working memory performance.
Time Frame: Baseline, 3-4 weeks
Population: 12 participants completed the n-back working memory task at both Baseline and Post-Testing, however one participant used an incorrect button to make responses at Baseline, so these responses were not recorded, leaving 11 participants with recorded data at Baseline and Post-Testing. Of these 11, 5 performed below chance (<50% hit rate) on the control task at one or both timepoints and were excluded from analysis.
Measure: Mean (Standard Deviation); unit: calculated score
Arm/Group | Experimental: HD-tDCS
Number analyzed (Participants) | 6
calculated score
  Baseline | 0.94 (0.72)
  3-4 weeks | 1.24 (0.60)
Statistical Analysis 1: Comparison: Experimental: HD-tDCS; Test type: Superiority; p = 0.168, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Experimental: HD-tDCS
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 13/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: HD-tDCS (N=13)
Progression of preexisting delusions related to Lewy Body Dementia disease progression (Nervous system disorders) | 1 — Changes of environment are known to be potential causes of worsening dementia symptoms. Participant was relocated to participate in the study.
Itching (Skin and subcutaneous tissue disorders) | 7
Worsening of dizziness upon standing post treatment (General disorders) | 1
Burning sensation (Skin and subcutaneous tissue disorders) | 13
Tingling (General disorders) | 13
Scalp Pain (Skin and subcutaneous tissue disorders) | 7
Trouble Concentrating (General disorders) | 5
Sleepiness (General disorders) | 8
Headache (General disorders) | 3
Acute Mood Change (General disorders) | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Skin Redness (Skin and subcutaneous tissue disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT04817891/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/91/NCT04817891/ICF_001.pdf